CLINICAL TRIAL: NCT05790707
Title: EfFect of Ablation of Persistent AtriaL Fibrillation on COgNitive Function in Individuals With Mild Cognitive Impairment : - The FALCON Study-
Brief Title: EfFect of Ablation of Persistent AtriaL Fibrillation on COgNitive Function in Individuals With Mild Cognitive Impairment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FALCON study
Record Dates: First submitted 2023-02-05; First posted 2023-03-30 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Mild Cognitive Impairment; Persistent Atrial Fibrillation
MeSH Terms: conditions — Cognitive Dysfunction; Atrial Fibrillation | interventions — Anti-Arrhythmia Agents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atrial fibrillation + antiarrhythmic drugs (Experimental): The ablation can be done with different sources of energy (radiofrequency, cryoballoon or pulsed field ablation). Different sets of lesions can be performed but the cornerstone is pulmonary vein isolation which will be mandatory.
  Antiarrhythmic drugs management will be at the operator discretion. Some operators may stop antiarrhythmic drugs after atrial fibrillation ablation.
  Interventions: Procedure: Atrial fibrillation ablation + antiarrhythmic drugs
- Antiarrhythmic drugs alone (Active Comparator): Antiarrhythmic drugs available available are amiodarone, flecainide, propafenone, sotalol.
  If not previously started, patients randomized to antiarrhythmic drugs arm should start antiarrhythmic drugs therapy within 1 week of randomization.
  Apart from these recommendations, antiarrhythmic drugs management will be at the operator discretion.
  Interventions: Drug: Antiarrhythmic drug

INTERVENTIONS:
Procedure: Atrial fibrillation ablation + antiarrhythmic drugs — Atrial fibrillation ablation will be performed with endovascular catheters and will be done either with radiofrequency, cryoballoon or pulsed field ablation.
  Amiodarone, flecainide, sotalol, propafenone are the anti arrhythmic drugs allowed.
  Arms: Atrial fibrillation + antiarrhythmic drugs
Drug: Antiarrhythmic drug — Amiodarone, flecainide, sotalol, propafenone are the anti arrhythmic drugs allowed.
  Arms: Antiarrhythmic drugs alone

SUMMARY:
The goal of this clinical trial is to evaluate the effect of catheter ablation of persistent atrial fibrillation on cognitive function in patients with mild cognitive impairment. Participants will be randomized into antiarrhythmic drugs alone or atrial fibrillation ablation + antiarrhythmic drugs.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 60 to 80 years
* Persistent atrial fibrillation
* Patients with an indication for cardiac rhythm control.
* Montreal Cognitive Assessment score between 18 and 25 points corresponding to mild cognitive impairment
* Free subject, not under temporary or permanent guardianship and not subject to subordination
* Subject understanding and accepting the constraints of the study
* Patient covered by French national health insurance or benefiting from it through a third party
* Subject has given written consent to the study after having received clear and complete information

Exclusion Criteria:

* Impossibility to perform the neuropsychological evaluation (communication problems such as hearing loss or aphasia, language barrier)
* History of clinical stroke
* Presence of a bruit at carotid auscultation or history of severe carotid stenosis
* History or suspicion of neurodegenerative disease (Parkinson's disease, Alzheimer's disease, Huntington's disease and amyotrophic lateral sclerosis...), bipolar disorder, schizophrenia, severe depression or amyloidosis
* Patient with history of previous atrial fibrillation ablation
* Patient undergoing flutter ablation or atrial tachycardia ablation (not atrial fibrillation ablation)
* Contraindication to atrial fibrillation ablation (intracardiac thrombus, severe pulmonary hypertension, mechanical mitral valve prosthesis or contraindication to anticoagulation,…)
* Contraindication to antiarrhythmic drugs, or to implantable cardiac monitor
* Patient with very advanced persistent atrial fibrillation, i.e., for more than 3 years or with a left atrial diameter >60 mm in parasternal long axis section or a left atrial volume > 48ml/m2 in echocardiography
* Subject with a life expectancy of less than 24 months at study enrolment
* Inability to consent
* Persons benefiting from a reinforced protection, namely minors, persons deprived of liberty by a judicial or administrative decision, adults under legal protection, and finally patients in emergency situations
* Pregnant or breastfeeding women, women at age to procreate and not using effective contraception (hormonal/barrier: oral, parenteral, percutaneous implantable, intrauterine device, or surgical: tubal ligation, hysterectomy, total ovariectomy)

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-04-21 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessmentquestionnaire score evolution 6 months | baseline (randomization) and 6 months after randomization
  To evaluate the effect of "atrial fibrillation ablation + antiarrhythmic drugs" on cognitive function as assessed by the change at the Montreal Cognitive Assessment questionnaire score between randomization (M0) and 6 months after randomization (M6), compared with "antiarrhythmic drugs alone" in patients with persistent atrial fibrillation associated with mild cognitive impairment. The Montreal Cognitive Assessment questionnaire score ranges from 0 to 30. A higher score indicates better cognitive performance.

SECONDARY OUTCOMES:
Baseline characteristics associated with Montreal Cognitive Assessment score improvement | baseline (randomization) and 6 months after randomization
  To define the baseline characteristics associated with Montreal Cognitive Assessment improvement between randomization (M0) and 6 months after randomization (M6) in patients with mild cognitive impairment and persistent atrial fibrillation undergoing atrial fibrillation ablation. The Montreal Cognitive Assessment questionnaire score ranges from 0 to 30. A higher score indicates better cognitive performance.
Changes in different types of cognitive functions | baseline (randomization) and 6 months after randomization
  To assess changes in different cognitive functions measured by a comprehensive neurocognitive assessment between randomization (M0) and 6 months after randomization (M6). The assessed tests are : Free recall/indexed recall 16, WAIS IV "digit memory" subtest, Rapid Frontal Efficiency Battery (BREF) score, Trail Making Test (TMT- GREFEX version), Verbal fluency (GREFEX version) categorical (animals) and literal (letter P), Oral naming of the BETL (Battery for the Evaluation of Language Disorders), STROOP test (GREFEX version), Rey figure, Processing speed index from the WAIS IV.
Montreal Cognitive Assessment questionnaire score evolution 12 months | baseline (randomization) and 12 months after randomization
  To evaluate the effect of "atrial fibrillation ablation + antiarrhythmic drugs" on cognitive function as assessed by the change at the Montreal Cognitive Assessment questionnaire score between randomization (M0) and 12 months after randomization (M12), compared with "antiarrhythmic drugs alone". The Montreal Cognitive Assessment questionnaire score ranges from 0 to 30. A higher score indicates better cognitive performance.
Association between atrial fibrillation burden and cognitive function | baseline (randomization) and 12 months after randomization
  To evaluate the association between atrial fibrillation burden and cognitive function as assessed by the change at the Montreal Cognitive Assessment questionnaire score between randomization (M0) and 12 months after randomization (M12). The Montreal Cognitive Assessment questionnaire score ranges from 0 to 30. A higher score indicates better cognitive performance.
Quality of life Short Form Survey (SF-12) | baseline (randomization), 6 and 12 months after randomization
  To evaluate the effect of "atrial fibrillation ablation + antiarrhythmic drugs" on quality of life assessed by the change at the 12-Item Short Form Survey (SF-12) between randomization (M0), 6 and 12 months after randomization (M6 and M12), compared with "antiarrhythmic drugs alone". Score ranges from 0 to 100, with higher scores indicating better physical and mental health functioning.
Quality of life QOL-AD | baseline (randomization), 6 and 12 months after randomization
  To evaluate the effect of "atrial fibrillation ablation + antiarrhythmic drugs" on quality of life assessed by the change at the Quality of life in Alzheimer's Disease (QOL-AD) questionnaire scores between randomization (M0), 6 and 12 months after randomization (M6 and M12), compared with "antiarrhythmic drugs alone". Score ranges from 13 to 52. The higher the score, the better quality of life the participant has.

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - CHU Angers, Angers
  - University Hospital, Brest
  - University Hospital, Caen
  - University Hospital, Dijon
  - CHU Grenoble, Grenoble
  - La Timone, Marseille
  - University Hospital, Poitiers
  - Centre Cardiologique du Nord, Saint-Denis